CLINICAL TRIAL: NCT03305133
Title: Evaluation of PD-L1 Tumor Expression in Patients With Large-cell Neuroendocrine Carcinoma (NEC) (EPNEC-GFPC 03-2017)
Brief Title: Evaluation of PD-L1 (Programmed Death-Ligand 1) Tumor Expression in Patients With Large-cell Neuroendocrine Carcinoma (NEC)
Acronym: EPNEC
Status: Completed | Type: Observational
Sponsor: Groupe Francais De Pneumo-Cancerologie (Other)
Responsible Party: Sponsor
Other Study IDs: GFPC 03-2017
Record Dates: First submitted 2017-10-04; First posted 2017-10-09 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Large Cell Lung Cancer; Neuroendocrine Carcinoma of Lung (Diagnosis)
MeSH Terms: conditions — Disease | interventions — Immunohistochemistry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Slides (tumour materials) at diagnosis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Immunohistochemistry — The slides which allowed the large cell neuroendocrine carcinoma diagnosis will be re-read centrally.

SUMMARY:
Observational, multicentre, retrospective study on patients taken care according to the national guidelines. The objective is to define, after the diagnosis confirmation, the frequency of PD-L1 expression in patients with large-cell lung neuroendocrine carcinoma (NEC), whatever the stage of the disease, and to correlate this parameter to clinical data at the time of diagnosis, therapeutic response and survival. Large-cell NECs present a bad prognostic and there is no evidence of treatment for these patients with advanced disease in second ligne of treatment at that time. To demonstrate the PD-L1 expression in this type of cancer might have a major therapeutic impact in a close future to access immunotherapies.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > or = 18 years
* Diagnosis of Large-cell NEC confirmed by centralised reading
* Tumoral materials available and readable for PD-L1 labeling

Exclusion Criteria:

* Other type of Lung cancers
* Tumoral material not available or not readable for centralised reading
* Tumoral material not available or not readable for PD-L1 labeling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting a large-cell NEC taken in charge by investigational centres between January 1st, 2014 and December 31st, 2016.
  Alive patients will be identified during disease follow-up visit as per the local current practice and the study will be then proposed to them at that time.
  For died patients, eligible patients will be identified by checking the files present at site by the Principal Investigator.
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Frequency of PD-L1 expression in patients with large-cell neuroendocrine carcinoma (NEC) | Retrospective central evaluation on tumour materials (slides) collected on patients diagnosed with NEC between 01 January 2014 and 31 December 2016
  Determine the frequency of PD-L1 expression in patients with large-cell neuroendocrine carcinoma (NEC)in terms of percentage of tumor cells expressing PD-L1 in immunohistochemistry (IHC) at the time of diagnosis:
  The frequency of PD-L1 expression determined by IHC will be as follow:
  * Negative PD-L1 tumours (<1% of positive tumour cells)
  * Positive PD-L1 tumours (> or = to 1% of positive tumour cells)
  * Low positive PD-L1 tumours (from 1% to 49% of positive tumour cells expressed)
  * High positive PD-L1 tumours (> or = 50% of positive tumour cells expressed)

SECONDARY OUTCOMES:
Correlation of PD-L1 expression of tumour cells with clinical data | Retrospective-data collected on patients diagnosed with NEC between 01 January 2014 and 31 December 2016
  Describe the disease at the time of diagnosis using TNM IASLC/UICC 2009 classification
Objective Response Rate (ORR) | Retrospective-data collected on patients diagnosed with NEC between 01 January 2014 and 31 December 2016
  Objective Response Rate (ORR): best overall response of complete response (CR) or partial response (PR) to a first line of treatment using RECIST 1.1 criteria as assessed locally
Progression-free survival (PFS) | Retrospective-data collected on patients diagnosed with NEC between 01 January 2014 and 31 December 2016
  PFS of the first line of treatment using RECIST 1.1 criteria assessed locally defined as the time from first treatment start to disease progression or death for any cause expressed in months
Overall survival (OS) | Retrospective-data collected on patients diagnosed with NEC between 01 January 2014 and 31 December 2016
  OS defined as the time from first treatment start to death for any cause expressed in months

CONTACTS AND LOCATIONS:
Overall Officials: Dominque Arpin, MD, Principal Investigator — Service de pneumologie et oncologie thoracique - Hôpital Nord-Ouest - F-69400 Villefranche sur Saône
Locations (28):
- France (28):
  - Centre Hospitalier D Argenteuil, Argenteuil, VAL D'oise
  - Site 12, Aix-en-Provence
  - Centre Hospitalier Universitaire, Angers
  - Site 05, Bastia
  - Site 22, Beauvais
  - Centre Hospitalier du Morvan, Brest
  - Site 43, Caen
  - Site 48, Clermont-Ferrand
  - Site 33, Créteil
  - Site 32, Elbeuf
  - Site 04, Gap
  - Centre Hospitalier Les Oudairies, La Roche-sur-Yon
  - Centre Hospitalier Universitaire DUPUYTREN, Limoges
  - Hospital du Cluzeau, Limoges
  - Site 00, Limoges
  - Centre Hospitalier Lyon Sud, Lyon
  - Site 25, Mantes-la-Jolie
  - Site 06, Marseille
  - Site 01, Meaux
  - Site 42, Orléans
  - Hospital Saint Antoine, Paris
  - Site 26, Paris
  - Site 19, Périgueux
  - Site 02, Reims
  - Site 18, Rouen
  - Site 17, Rouen
  - Site 14, Toulon
  - Site 11, Villefranche-sur-Saône

IPD SHARING:
Plan to Share IPD: Undecided